CLINICAL TRIAL: NCT06929715
Title: Effect of an Educational Intervention on CPR Knowledge and Skills in 7- and 8-Year-Old Schoolchildren: A Non-Randomized Controlled Trial
Brief Title: Effect of an Educational Intervention on CPR Knowledge and Skills in Schoolchildren
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Responsible Party: Principal Investigator, Diana Maria Blanco Avila, Principal researcher, Universidad Nacional de Colombia
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AVAL 20-24; AVAL 20-24 (Other: Universidad Nacional de Colombia)
Record Dates: First submitted 2025-03-20; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: CPR; Cardiac Arrest (CA)
Keywords: schoolchildren; learning; intervention; knowledge; skills
MeSH Terms: conditions — Heart Arrest | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: In this study, masking is implemented to minimize bias in outcome assessment. Specifically, both the participants and the investigators conducting the measurements are blinded to the group assignments. In addition, the statistician responsible for data analysis remains masked to the intervention allocation. To further reduce potential contamination, different educational institutions have been selected for each arm of the study. This comprehensive masking approach ensures that data collection, evaluation, and analysis are conducted without bias from knowledge of group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): This group of students receives the structured educational program designed to teach the first link in the chain of survival, specifically tailored for their age. The intervention is delivered in the school setting and focuses on enhancing the knowledge and practical CPR skills of 7- and 8-year-old children.
  Interventions: Other: Intervention for Teaching the First Link in the Chain of Survival to 7- and 8-Year-Old Children
- Control Arm (Placebo Comparator): This group does not receive the CPR educational intervention during the study period but will receive a first aid intervention that does not include teaching the first link in the chain of survival. This group serves as a reference to compare and evaluate the effectiveness of the program implemented in the intervention group.
  Interventions: Other: Placebo Intervention - First Aid (Excluding Basic CPR)

INTERVENTIONS:
Other: Intervention for Teaching the First Link in the Chain of Survival to 7- and 8-Year-Old Children — Unlike traditional CPR training programs designed primarily for older children or adults, this intervention is uniquely tailored for 7- and 8-year-old schoolchildren. It employs a narrative-based, age-appropriate educational approach that incorporates storytelling, interactive activities, and practical simulation exercises aligned with the cognitive and motor development of young learners. Delivered by school nurses in a classroom setting, the program not only focuses on teaching the first link in the chain of survival but also ensures that its content and methods are rigorously validated by experts. Moreover, the intervention includes a follow-up evaluation at three months to assess the retention of knowledge and skills, distinguishing it from other clinical studies that lack such long-term assessment.
  Arms: Intervention Arm
Other: Placebo Intervention - First Aid (Excluding Basic CPR) — In the control arm, participants receive a structured first aid educational program that intentionally excludes any training on the first link in the chain of survival. This intervention focuses on general first aid skills-such as wound care, management of minor injuries, and other non-cardiac emergency procedures-ensuring that no content related to recognizing a cardiac emergency or activating the emergency response system is provided. Delivered in a classroom setting by qualified personnel, the program is designed to mirror the overall structure, duration, and engagement level of the CPR intervention without overlapping its core content. Expert validation has been obtained to confirm that the curriculum remains neutral and strictly adheres to general first aid, thereby serving as a robust comparator to isolate the specific effects of CPR training in young schoolchildren.
  Arms: Control Arm

SUMMARY:
This study aims to evaluate the effectiveness of a CPR intervention for children aged 7 and 8. Given the high prevalence of out-of-hospital cardiac arrests (OHCA) and the proven benefits of early CPR training, the study seeks to determine whether a structured intervention can improve young children's knowledge and skills in basic life support.

What is the effect of a CPR training intervention on the knowledge and skills of 7- and 8-year-old schoolchildren?

Cardiac arrest is a leading cause of mortality worldwide. Research shows that survival rates increase significantly when CPR is performed promptly by a trained bystander. Countries with early CPR training programs in schools, such as Norway and Denmark, report better survival outcomes. However, in Latin America, CPR education in schools is still in its early stages. Evidence suggests that children can effectively learn and retain CPR knowledge, and they can serve as multipliers by passing their knowledge to family and peers.

Study Design:

This is a non-randomized, double-blind controlled trial with four phases:

DETAILED DESCRIPTION:
Intervention Design - Developing an age-appropriate CPR training intervention based on educational and cognitive development theories.

Content Validation - Experts in child education and health professionals will assess the content and delivery methods.

Validation of Assessment Tools - Ensuring reliability in measuring children's CPR knowledge and skills.

Intervention Implementation and Evaluation - The intervention will be conducted in schools, with pre- and post-tests assessing knowledge and skills retention after 3 months.

Expected Outcomes:

Improved knowledge and skill levels in CPR among children who receive the intervention.

Validation of a structured educational approach for teaching CPR to young children.

Contribution to global evidence on CPR education and its potential impact in Bogotá schools.

ELIGIBILITY:
Inclusion Criteria:

* Schoolchildren aged between 7 and 8 years.
* Students enrolled in an educational institution that has authorized their participation in the study.
* Not participating in any other intervention or educational program related to CPR during the study period.

Exclusion Criteria:

* Students whose parents, legal guardians, teachers, or the students themselves report any health condition that prevents them from participating in the study.
* Students who indicate having received prior training in CPR or related skills.
* Students whose parents, legal guardians, or teachers report any cognitive condition that limits their ability to understand and follow the instructions necessary to learn and practice CPR in simulated scenarios.

Ages: 7 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 388 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in knowledge and practical skills in basic CPR-specifically, the first link in the chain of survival | 3 moths
  The primary outcome measure for this study is the change in knowledge and practical skills in basic CPR-specifically, the first link in the chain of survival-among 7- and 8-year-old schoolchildren. This will be assessed through a structured pre- and post-intervention questionnaire that evaluates theoretical understanding of CPR and an observational checklist used during simulated scenarios to gauge practical skill execution.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Nacional de Colombia, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pedrazas-Lopez D, de Pablo-Marquez B, Cunillera-Puertolas O, Almeda-Ortega J; Grupo de Investigacion RCParvulari. RCParvulari training: A basic life support training methodology applied to 5-year-old students: Effectiveness in a cluster-randomized clinical trail. An Pediatr (Engl Ed). 2023 Feb;98(2):99-108. doi: 10.1016/j.anpede.2023.01.006. Epub 2023 Feb 3. PMID 36740509
- [Background] Nakagawa NK, Salles IC, Semeraro F, Bottiger BW. KIDS SAVE LIVES: a narrative review of associated scientific production. Curr Opin Crit Care. 2021 Dec 1;27(6):623-636. doi: 10.1097/MCC.0000000000000872. PMID 34495875
- [Background] Navarro-Paton R, Freire-Tellado M, Fernandez-Gonzalez N, Basanta-Camino S, Mateos-Lorenzo J, Lago-Ballesteros J. What is the best position to place and re-evaluate an unconscious but normally breathing victim? A randomised controlled human simulation trial on children. Resuscitation. 2019 Jan;134:104-109. doi: 10.1016/j.resuscitation.2018.10.030. Epub 2018 Oct 30. PMID 30389590
- [Background] Stroobants J, Monsieurs K, Devriendt B, Dreezen C, Vets P, Mols P. Schoolchildren as BLS instructors for relatives and friends: Impact on attitude towards bystander CPR. Resuscitation. 2014 Dec;85(12):1769-74. doi: 10.1016/j.resuscitation.2014.10.013. PMID 25447432
- [Background] Ong ME, Shin SD, De Souza NN, Tanaka H, Nishiuchi T, Song KJ, Ko PC, Leong BS, Khunkhlai N, Naroo GY, Sarah AK, Ng YY, Li WY, Ma MH; PAROS Clinical Research Network. Outcomes for out-of-hospital cardiac arrests across 7 countries in Asia: The Pan Asian Resuscitation Outcomes Study (PAROS). Resuscitation. 2015 Nov;96:100-8. doi: 10.1016/j.resuscitation.2015.07.026. Epub 2015 Jul 30. PMID 26234891
- [Background] De Buck E, Van Remoortel H, Dieltjens T, Verstraeten H, Clarysse M, Moens O, Vandekerckhove P. Evidence-based educational pathway for the integration of first aid training in school curricula. Resuscitation. 2015 Sep;94:8-22. doi: 10.1016/j.resuscitation.2015.06.008. Epub 2015 Jun 18. PMID 26093230
- [Background] Suss-Havemann C, Kosan J, Seibold T, Dibbern NM, Daubmann A, Kubitz JC, Beck S. Implementation of Basic Life Support training in schools: a randomised controlled trial evaluating self-regulated learning as alternative training concept. BMC Public Health. 2020 Jan 13;20(1):50. doi: 10.1186/s12889-020-8161-7. PMID 31931770
- [Background] Yeung J, Kovic I, Vidacic M, Skilton E, Higgins D, Melody T, Lockey A. The school Lifesavers study-A randomised controlled trial comparing the impact of Lifesaver only, face-to-face training only, and Lifesaver with face-to-face training on CPR knowledge, skills and attitudes in UK school children. Resuscitation. 2017 Nov;120:138-145. doi: 10.1016/j.resuscitation.2017.08.010. Epub 2017 Oct 1. PMID 28974344
- [Background] Bohn A, Van Aken H, Lukas RP, Weber T, Breckwoldt J. Schoolchildren as lifesavers in Europe - training in cardiopulmonary resuscitation for children. Best Pract Res Clin Anaesthesiol. 2013 Sep;27(3):387-96. doi: 10.1016/j.bpa.2013.07.002. PMID 24054517
- [Background] Universidad Nacional de Colombia - Sede Bogotá, Enfermería F de. Avances de investigación en la Facultad de Enfermería. Editorial. Vol. 1, Editorial Universidad Nacional de Colombia. 2022. 1-426 p.
- [Background] Malta Hansen C, Kragholm K, Pearson DA, Tyson C, Monk L, Myers B, Nelson D, Dupre ME, Fosbol EL, Jollis JG, Strauss B, Anderson ML, McNally B, Granger CB. Association of Bystander and First-Responder Intervention With Survival After Out-of-Hospital Cardiac Arrest in North Carolina, 2010-2013. JAMA. 2015 Jul 21;314(3):255-64. doi: 10.1001/jama.2015.7938. PMID 26197186
- [Background] Wissenberg M, Lippert FK, Folke F, Weeke P, Hansen CM, Christensen EF, Jans H, Hansen PA, Lang-Jensen T, Olesen JB, Lindhardsen J, Fosbol EL, Nielsen SL, Gislason GH, Kober L, Torp-Pedersen C. Association of national initiatives to improve cardiac arrest management with rates of bystander intervention and patient survival after out-of-hospital cardiac arrest. JAMA. 2013 Oct 2;310(13):1377-84. doi: 10.1001/jama.2013.278483. PMID 24084923
- [Background] Plant N, Taylor K. How best to teach CPR to schoolchildren: a systematic review. Resuscitation. 2013 Apr;84(4):415-21. doi: 10.1016/j.resuscitation.2012.12.008. Epub 2012 Dec 11. PMID 23246989
- [Background] Bottiger BW, Lockey A, Aickin R, Castren M, de Caen A, Escalante R, Kern KB, Lim SH, Nadkarni V, Neumar RW, Nolan JP, Stanton D, Wang TL, Perkins GD. "All citizens of the world can save a life" - The World Restart a Heart (WRAH) initiative starts in 2018. Resuscitation. 2018 Jul;128:188-190. doi: 10.1016/j.resuscitation.2018.04.015. Epub 2018 Apr 19. PMID 29679697
- [Background] Semeraro F, Greif R, Bottiger BW, Burkart R, Cimpoesu D, Georgiou M, Yeung J, Lippert F, S Lockey A, Olasveengen TM, Ristagno G, Schlieber J, Schnaubelt S, Scapigliati A, G Monsieurs K. European Resuscitation Council Guidelines 2021: Systems saving lives. Resuscitation. 2021 Apr;161:80-97. doi: 10.1016/j.resuscitation.2021.02.008. Epub 2021 Mar 24. PMID 33773834